CLINICAL TRIAL: NCT00537290
Title: A Pilot Study of Rituximab for the Anticoagulation Resistant Manifestations of Antiphospholipid Syndrome (RITAPS)
Brief Title: A Pilot Study of Rituximab for the Anticoagulation Resistant Manifestations of Antiphospholipid Syndrome
Acronym: RITAPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 27022
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Antiphospholipid Syndrome
Keywords: antiphospholipid syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): All patients will receive 1000 milligrams of rituximab by intravenous infusion on Days 1 and 15.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000mg IV on Days 0 and 15
  Other Names: Rituxan

SUMMARY:
RITuximab AntiphosPholipid Syndrome (RITAPS) Study is designed to evaluate whether a medication called rituximab would reduce the signs and symptoms of antiphospholipid antibody (aPL) -related certain clinical problems.

DETAILED DESCRIPTION:
Persistently antiphospholipid antibody (aPL)-positive patients, age 18 - 75 years of age, with anticoagulation-resistant manifestations of APS and fulfilling protocol defined study inclusion criteria will receive two doses of Rituximab, and will be followed for 6 and 12 months for clinical and safety outcomes, respectively.

Patients are eligible to take part in this study if their blood test is persistently positive for aPL and they have one or more of the aPL-related clinical problem(s) listed below: low platelet (blood cells involved in the prevention of bleeding) count; anemia (deficiency of red blood cells); heart valve disease; skin ulcers; kidney smal vessel blood clots; and/or memory problems.

ELIGIBILITY:
Inclusion Criteria:

* - Positive aPL profile defined as:

  * Positive lupus anticoagulant test as defined by the International Society on Thrombosis and Haemostasis, on two or more occasions, at least 12 weeks apart and/or
  * Positive anticardiolipin antibody (aCL) immunoglobulin G(Ig)G/M/A isotype, present in > 40U, on two or more occasions, at least 12 weeks apart and/or
  * Positive anti-β2-glycoprotein-I (aβ2GPI) IgG/M/A isotype, present in > 40U, on two or more occasions, at least 12 weeks apart

AND

- Clinical features attributable to aPL that are resistant to warfarin and/or heparin:

* Persistent thrombocytopenia and/or
* Persistent autoimmune hemolytic anemia and/or
* Cardiac valve disease and/or
* Chronic skin ulcers and/or
* Renal thrombotic microangiopathy and/or
* Cognitive dysfunction with/without white matter changes

Exclusion Criteria (selected):

* > 4/11 American College of Rheumatology Classification Criteria for SLE
* Acute thrombosis
* History of stroke (only for patients with cognitive dysfunction)
* Positive Hepatitis B or C serology
* History of positive HIV
* Acute or chronic pancreatitis
* Treatment with any investigational agent within 4 weeks of screening
* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab (MabThera® / Rituxan®)
* Previous treatment with Natalizumab (Tysabri®)
* Known active bacterial, viral fungal mycobacterial, or other infection
* Pregnancy
* Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder that would interfere with normal participation in this protocol
* Significant cardiac or pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doruk Erkan, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Barbara Volcker Center for Women and Rheumatic Disease, Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erkan D, Vega J, Ramon G, Kozora E, Lockshin MD. A pilot open-label phase II trial of rituximab for non-criteria manifestations of antiphospholipid syndrome. Arthritis Rheum. 2013 Feb;65(2):464-71. doi: 10.1002/art.37759. PMID 23124321
- [Derived] Khattri S, Zandman-Goddard G, Peeva E. B-cell directed therapies in antiphospholipid antibody syndrome--new directions based on murine and human data. Autoimmun Rev. 2012 Aug;11(10):717-22. doi: 10.1016/j.autrev.2011.12.011. Epub 2012 Jan 16. PMID 22269862
- See also: Hospital for Special Surgery Clinical Trials List — http://www.hss.edu/clinical-trials-directory.asp
- See also: Barbara Volcker Center for Women and Rheumatic Disease — http://www.hss.edu/barbara-volcker.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were ≥18 years of age, did not have other systemic autoimmune diseases, and fulfilled at least one of the laboratory criteria and one of the clinical criteria were eligible for inclusion in the study.
Pre-assignment Details: Laboratory criteria defined as positive results of a LAC test, positive aCL IgG/IgM/IgA isotype (≥40), and/or positive anti-β2GPI IgG/IgM/IgA isotype (≥40) on 2 or more occasions, at least 12 weeks apart. Clinical criteria defined as 1)persistent thrombocytopenia 2)Cardiovascular disease 3)skin ulcer 4)aPL nephropathy 5) cognitive dysfunction.
Period: Overall Study
Arm/Group | Rituximab
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients included in the study
Arm/Group | Rituximab
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — The mean age of the patients
  years | 40.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution
  Participants
    Female | 11
    Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race distribution
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 17
    More than one race | 0
    Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants] — Region of the patients
  Participants
    United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Serious and Non Serious Adverse Events
Description: Serious and non-serious adverse events were evaluated throughout 52 weeks + additional 4 months for the patients with low B cell counts.
Time Frame: 52 weeks + additional 4 months if needed
Population: All patients enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: The Efficacy of Rituximab
Description: Outcome measures scored as complete response(CR),partial(PR),and none(NR) at 24 weeks.For thrombocytopenia,CR defined as a platelet count of ≥150×109/μl,PR as 100-149,and NR as <100.For CVD,CR defined as the disappearance of cardiac lesions,PR as 50%improvement,and NR as no change.For skin ulcer,CR defined as disappearance,PR as 50% improvement,and NR as no change.For aPL nephropathy,CR defined as a normal serum creatinine level,inactive urinary sediment,and urinary protein:creatinine 0.5;PR as a serum cr level 15%above baseline,RBCs per high-power field 50%above baseline with no casts,50%improvement in the urinary prt:cr,and estimated GFR 10%above baseline;and NR as the absence of C/PR.For cognitive dysfunction,CR defined as normalization of the cognitive impairment index with 50%improvement,PR as abnormal index with 50%,and NR as no change.
Time Frame: 24 weeks
Population: All patients enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 19
Participants
  Complete Response | 7
  Partial Response | 4
  No Response | 6
  Could not tolerate the infusion (not evaluated) | 2

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality. A serious adverse event (SAE) was defined as an AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=19)
Antiepileptic drug adjustment (history of seizure disorder) (Nervous system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Brain surgery (history of seizure disorder) (Nervous system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Subdural hematoma (Nervous system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
New-onset focal motor seizure due to previous stroke (Nervous system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
48-hour EEG monitoring and new-onset partial sensory seizure (Nervous system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Pneumonia (Infections and infestations) | 2 (2) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Viral gastroenteritis/dehydration/cellulitis (Infections and infestations) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Recurrent deep vein thrombosis (Vascular disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Post-phlebitic syndrome (Vascular disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Multifocal atrial tachycardia due to resolving pneumonia (Cardiac disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
Allergy-Trimethoprim/sulfamethoxazole treatment (Immune system disorders) | 1 (1) — A serious adverse event (SAE) was defined as an adverse event AE meeting ≥1 of the following criteria: death, life-threatening, requiring or prolonging inpatient hospitalization, disabling, or resulting in a congenital anomaly.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=19)
Chest pain with fever, chills, and low back pain (Cardiac disorders) | 1 (2) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Transient chest pressure (Cardiac disorders) | 3 (3) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Diffuse severe erythematous rash (Skin and subcutaneous tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Facial rash (Skin and subcutaneous tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Nausea (Gastrointestinal disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Transient palpitations (recurrence) (Cardiac disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Deep vein thrombosis (recurrence) (Vascular disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Raynaud's phenomenon (new) (Vascular disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Rash (diffuse) within 1 week of rituximab infusion (new) (Skin and subcutaneous tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Rash (local) within 1 week of rituximab infusion (new) (Skin and subcutaneous tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Rash (local) due to nail glue allergy (new) (Skin and subcutaneous tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Gastrointestinal reflux disease (new) (Gastrointestinal disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Epistaxis (recurrence) (Blood and lymphatic system disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Upper respiratory tract infection (Infections and infestations) | 6 (6) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Tonsillitis, otitis, sinusitis (Infections and infestations) | 3 (3) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Urinary tract infection (Infections and infestations) | 3 (3) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Bronchitis (Infections and infestations) | 2 (2) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Acute gastroenteritis (Infections and infestations) | 2 (2) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Cellulitis (Infections and infestations) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Herpes zoster infection within 2 weeks of rituximab infusion (new) (Infections and infestations) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Herpes zoster infection while noncompliant with prophylaxis (recurrence) (Infections and infestations) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Arthralgia (local) (new) (Musculoskeletal and connective tissue disorders) | 2 (2) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Arthritis (diffuse) within 1 week of the infusion (new) (Musculoskeletal and connective tissue disorders) | 2 (2) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Arthralgia (diffuse) within 2 weeks of the infusion (new) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Arthralgia (local) (recurrence) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Carpal tunnel syndrome (recurrence) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Gout flare (recurrence) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Shoulder dislocation (new) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Elbow incidental MRI metallic artifact finding (new) (Musculoskeletal and connective tissue disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Seizures (history of partially controlled seizures) (recurrence) (Nervous system disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Depression (new) (Psychiatric disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Migraine (new) (Nervous system disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.
Headache (severe, transient) (new) (Nervous system disorders) | 1 (1) — An adverse event (AE) was defined as any unfavorable medical occurrence, regardless of causality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No